CLINICAL TRIAL: NCT04559568
Title: A Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study of Single- and Multiple-Ascending Doses of LY3522348 in Healthy Participants
Brief Title: A Study of LY3522348 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 17808; J2U-MC-YBAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-09-21; First posted 2020-09-23 (Actual); Results first posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Part A: Placebo (Placebo Comparator): A single dose of Placebo administered orally on Day 1.
  Interventions: Drug: Placebo
- Part A: 5 milligrams (mg) LY3522348 (Experimental): A single dose of 5 mg LY3522348 administered orally on Day 1.
  Interventions: Drug: LY3522348
- Part A: 15 mg LY3522348 (Experimental): A single dose of 15 mg LY3522348 administered orally on Day 1.
  Interventions: Drug: LY3522348
- Part A: 50 mg LY3522348 (Experimental): A single dose of 50 mg LY3522348 administered orally on Day 1.
  Interventions: Drug: LY3522348
- Part A: 150 mg LY3522348 (Experimental): A single dose of 150 mg LY3522348 administered orally on Day 1.
  Interventions: Drug: LY3522348
- Part A: 380 mg LY3522348 (Experimental): A single dose of 380 mg LY3522348 administered orally on Day 1.
  Interventions: Drug: LY3522348
- Part B: Placebo (Placebo Comparator): Placebo administered orally once daily on Days 1-14.
  Interventions: Drug: Placebo
- Part B: Placebo + Midazolam (Experimental): Placebo administered orally once daily on Days 1-15 and a single dose of 200 micrograms (μg) Midazolam administered orally on Days -1 and 15.
  Interventions: Drug: Placebo; Drug: Midazolam
- Part B: 50 mg LY3522348 (Experimental): 50 mg LY3522348 administered orally once daily on Days 1-14.
  Interventions: Drug: LY3522348
- Part B: 120 mg LY3522348 (Experimental): 120 mg LY3522348 administered orally once daily on Days 1-14.
  Interventions: Drug: LY3522348
- Part B: 290 mg LY3522348 + Midazolam (Experimental): 290 mg LY3522348 administered orally once daily on Days 1-15 and a single dose of 200 μg Midazolam administered orally on Days -1 and 15.
  Interventions: Drug: LY3522348; Drug: Midazolam

INTERVENTIONS:
Drug: LY3522348 — Administered orally.
  Arms: Part A: 15 mg LY3522348; Part A: 150 mg LY3522348; Part A: 380 mg LY3522348; Part A: 5 milligrams (mg) LY3522348; Part A: 50 mg LY3522348; Part B: 120 mg LY3522348; Part B: 290 mg LY3522348 + Midazolam; Part B: 50 mg LY3522348
Drug: Placebo — Administered orally.
  Arms: Part A: Placebo; Part B: Placebo; Part B: Placebo + Midazolam
Drug: Midazolam — Administered orally.
  Arms: Part B: 290 mg LY3522348 + Midazolam; Part B: Placebo + Midazolam

SUMMARY:
The main purpose of this study in healthy participants is to learn more about the safety of LY3522348 and any side effects that might be associated with it. Blood tests will be performed to check how much LY3522348 gets into the bloodstream and how long it takes the body to eliminate it. This study has two parts: Part A will last up to about six weeks and Part B will last up to about eight weeks for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined through medical evaluation including medical history and physical examination
* Have a body mass index of greater than or equal to (≥)18.5 and less than or equal to (≤)40 kilograms per square meter (kg/m²)
* Have had a stable weight for one month prior to screening and enrollment (less than [<]5 percent [%] body weight change) and have not received dietary intervention in the one month prior to screening and enrollment
* Have safety laboratory test results within normal reference range for the population or investigative site, or results with acceptable deviations that are judged to be not clinically significant by the investigator

Exclusion Criteria:

* Have an abnormality in the 12-lead electrocardiogram (ECG) at screening that, in the opinion of the investigator, increases the risks associated with participating in the study or may confound ECG data analysis
* Have blood pressure of greater than (>)160/90 millimeters of mercury (mmHg) and pulse rate <50 or >100 beats per minute (bpm), supine (at screening), or with minor deviations judged to be acceptable by the investigator
* Have a history of fructosuria
* Use of any drugs or substances that are known strong inducers or inhibitors of cytochrome P450 3A4 (CYP3A) is specifically excluded within 14 days prior to the first administration of study intervention and during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Inc, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fukuda T, Thompson BR, Brouwers B, Qian HR, Wang W, Morse BL, LaBell ES, Durham TB, Konig M, Haupt A, Benson CT, MacKrell J. LY3522348, A New Ketohexokinase Inhibitor: A First-in-Human Study in Healthy Adults. Diabetes Ther. 2025 Jul;16(7):1399-1415. doi: 10.1007/s13300-025-01752-5. Epub 2025 May 13. PMID 40358849

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: 5 mg LY3522348: A single dose of 5 mg LY3522348 administered orally on Day 1.
- Part B: Placebo + Midazolam: Placebo administered orally once daily on Days 1-15 and a single dose of 200 μg Midazolam administered orally on Days -1 and 15.
Period: Overall Study
Arm/Group | Part A: Placebo | Part A: 5 mg LY3522348 | Part A: 15 mg LY3522348 | Part A: 50 mg LY3522348 | Part A: 150 mg LY3522348 | Part A: 380 mg LY3522348 | Part B: Placebo | Part B: Placebo + Midazolam | Part B: 50 mg LY3522348 | Part B: 120 mg LY3522348 | Part B: 290 mg LY3522348 + Midazolam
Started | 10 | 6 | 6 | 6 | 6 | 6 | 4 | 2 | 6 | 6 | 7
Received At Least 1 Dose of Study Drug | 10 | 6 | 6 | 6 | 6 | 6 | 4 | 2 | 6 | 6 | 7
Completed | 10 | 6 | 6 | 6 | 6 | 6 | 4 | 2 | 6 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Placebo | Part A: 5 mg LY3522348 | Part A: 15 mg LY3522348 | Part A: 50 mg LY3522348 | Part A: 150 mg LY3522348 | Part A: 380 mg LY3522348 | Part B: Placebo | Part B: Placebo + Midazolam | Part B: 50 mg LY3522348 | Part B: 120 mg LY3522348 | Part B: 290 mg LY3522348 + Midazolam | Total
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 4 | 2 | 6 | 6 | 7 | 65
Age, Continuous [Mean (Full Range); unit: years] | 50.2 [28 to 62] | 53.5 [43 to 64] | 48.8 [36 to 64] | 56.0 [38 to 65] | 57.0 [45 to 64] | 31.0 [27 to 36] | 47.5 [36 to 62] | 57.0 [55 to 59] | 43.0 [28 to 54] | 36.3 [29 to 39] | 45.0 [32 to 64] | 47.3 [27 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 5 | 3 | 4 | 0 | 2 | 1 | 2 | 1 | 1 | 26
  Male | 7 | 2 | 1 | 3 | 2 | 6 | 2 | 1 | 4 | 5 | 6 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 2 | 1 | 2 | 4 | 3 | 1 | 4 | 1 | 1 | 23
  Not Hispanic or Latino | 8 | 4 | 4 | 5 | 4 | 2 | 1 | 1 | 2 | 5 | 6 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 1 | 3 | 1 | 2 | 2 | 1 | 1 | 2 | 4 | 4 | 26
  White | 5 | 5 | 3 | 5 | 4 | 4 | 3 | 1 | 4 | 2 | 3 | 39
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: An SAE is any untoward medical occurrence temporally associated with the use of study intervention that results in death is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation as determined by investigator. The number of participants with one or more SAEs considered by the investigator to be related to study drug administration is reported here. A summary of SAEs and other non-serious adverse events, regardless of causality, will be reported in the Reported Adverse Events module.
Time Frame: Part A: Baseline up to Day 14; Part B: Baseline up to Day 28
Population: All enrolled participants, irrespective of the completion of all protocol requirements.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: 5 mg LY3522348 | Part A: 15 mg LY3522348 | Part A: 50 mg LY3522348 | Part A: 150 mg LY3522348 | Part A: 380 mg LY3522348 | Part B: Placebo | Part B: Placebo + Midazolam | Part B: 50 mg LY3522348 | Part B: 120 mg LY3522348 | Part B: 290 mg LY3522348 + Midazolam
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 4 | 2 | 6 | 6 | 7
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Part A Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to the Last Time Point With a Measurable Concentration (AUC(0-tlast)) of LY3522348
Description: PK: AUC(0-tlast) of LY3522348
Time Frame: Day 1 (Predose, 0.75, 1.5, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 144 hours post Day 1 dose)
Population: All enrolled participants in Part A who received at least one dose of study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour/milliliter (μg*h/mL)
Arm/Group | Part A: 5 mg LY3522348 | Part A: 15 mg LY3522348 | Part A: 50 mg LY3522348 | Part A: 150 mg LY3522348 | Part A: 380 mg LY3522348
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
microgram*hour/milliliter (μg*h/mL) | 0.330 (25) | 1.27 (30) | 3.37 (20) | 9.45 (37) | 25.3 (24)

3. Secondary Outcome: Part B PK: Area Under the Concentration Versus Time Curve From Time Zero to the Last Time Point With a Measurable Concentration (AUC(0-tlast)) of LY3522348
Description: PK: AUC(0-tlast) of LY3522348
Time Frame: Day 1 (Predose, 0.75, 1.5, 3, 4, 6, 8, 12, 16, 24 hours post Day 1 dose); Day 14 (Predose, 0.75, 1.5, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96, 144 hours post Day 14 dose)
Population: All enrolled participants in Part B who received at least one dose of study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | Part B: 50 mg LY3522348 | Part B: 120 mg LY3522348 | Part B: 290 mg LY3522348 + Midazolam
Number analyzed (Participants) | 6 | 6 | 6
μg*h/mL
  Day 1 | 1.76 (25) | 5.03 (18) | 11.1 (25)
  Day 14: number analyzed (Participants) | 6 | 5 | 6
  Day 14 | 6.00 (29) | 14.4 (31) | 20.4 (22)

4. Secondary Outcome: Part A PK: Maximum Observed Drug Concentration (Cmax) of LY3522348
Description: PK: Cmax of LY3522348
Time Frame: Day 1 (Predose, 0.75, 1.5, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 144 hours post Day 1 dose)
Population: All enrolled participants in Part A who received at least one dose of study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/mililiter (μg/mL)
Arm/Group | Part A: 5 mg LY3522348 | Part A: 15 mg LY3522348 | Part A: 50 mg LY3522348 | Part A: 150 mg LY3522348 | Part A: 380 mg LY3522348
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
micrograms/mililiter (μg/mL) | 0.00964 (17) | 0.0399 (23) | 0.113 (23) | 0.323 (39) | 0.897 (18)

5. Secondary Outcome: Part B PK: Maximum Observed Drug Concentration (Cmax) of LY3522348
Description: PK: Cmax of LY3522348
Time Frame: as for outcome 3
Population: All enrolled participants in Part B who received at least one dose of study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part B: 50 mg LY3522348 | Part B: 120 mg LY3522348 | Part B: 290 mg LY3522348 + Midazolam
Number analyzed (Participants) | 6 | 6 | 6
μg/mL
  Day 1 | 0.109 (29) | 0.330 (15) | 0.690 (13)
  Day 14: number analyzed (Participants) | 6 | 5 | 6
  Day 14 | 0.188 (25) | 0.464 (15) | 1.15 (22)

ADVERSE EVENTS:
Time Frame: Part A: Baseline up to Day 14; Part B: Baseline up to Day 28
Description: All enrolled participants, irrespective of the completion of all protocol requirements.
Arm/Group | Part A: Placebo | Part A: 5 mg LY3522348 | Part A: 15 mg LY3522348 | Part A: 50 mg LY3522348 | Part A: 150 mg LY3522348 | Part A: 380 mg LY3522348 | Part B: Placebo | Part B: Placebo + Midazolam | Part B: 50 mg LY3522348 | Part B: 120 mg LY3522348 | Part B: 290 mg LY3522348 + Midazolam
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/4 | 0/2 | 0/6 | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/4 | 0/2 | 0/6 | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 1/10 | 2/6 | 1/6 | 1/6 | 3/6 | 1/6 | 0/4 | 0/2 | 0/6 | 3/6 | 1/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Placebo (N=10) | Part A: 5 mg LY3522348 (N=6) | Part A: 15 mg LY3522348 (N=6) | Part A: 50 mg LY3522348 (N=6) | Part A: 150 mg LY3522348 (N=6) | Part A: 380 mg LY3522348 (N=6) | Part B: Placebo (N=4) | Part B: Placebo + Midazolam (N=2) | Part B: 50 mg LY3522348 (N=6) | Part B: 120 mg LY3522348 (N=6) | Part B: 290 mg LY3522348 + Midazolam (N=7)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site dermatitis (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asymptomatic COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/68/NCT04559568/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-03): https://cdn.clinicaltrials.gov/large-docs/68/NCT04559568/SAP_001.pdf